CLINICAL TRIAL: NCT02475707
Title: Administration of Donor-Derived Multi-Tumor-Associated Antigen (TAA)-Specific T Cells to Patients With ALL
Brief Title: Administration of Donor MultiTAA-Specific T Cells for ALL
Acronym: STELLA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Bilal Omer, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-37042 STELLA; STELLA (Other: Baylor College of Medicine)
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Leukemia, Lymphoblastic (Acute)
Keywords: leukemia; lymphoblastic; ALL; multiTAA-specific T cells; HSCT
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Treatment with donor-derived multiTAA-specific T cells as adjuvant therapy following HSCT for ALL.
  Interventions: Biological: MultiTAA-specific T cells
- Group B (Experimental): Treatment with donor-derived multiTAA-specific T cells for relapsed/residual disease following HSCT for ALL.
  Interventions: Biological: MultiTAA-specific T cells

INTERVENTIONS:
Biological: MultiTAA-specific T cells — The 3 dose levels are:
  Dose Level 1: 5 x 10e6 cells/m2; Dose Level 2: 1 x 10e7 cells/m2; Dose Level 3: 2 x 10e7 cells/m2
  The T cells are given from 30 days post-HSCT. They are administered by intravenous injection over 1-10 minutes through either a peripheral or a central line.
  Patients being treated on Arm A (adjuvant) or Arm B (active disease) who have a partial response, complete response or stable disease, will be eligible to receive up to 6 further doses of multiTAA-specific T cells at the same dose as the initial infusions at a minimum of 4 weeks apart.
  Other Names: Multiple tumor-associated antigen (TAA)-specific T cells

SUMMARY:
This study uses special blood cells called multiple tumor-associated antigen (TAA)-specific T cells to treat patients with acute lymphoblastic leukemia (ALL) which has come back, or may come back, or has not gone away after standard treatment, including an allogeneic hematopoietic stem cell transplant (HSCT).

The investigators have previously used this sort of therapy to treat Hodgkin or non-Hodgkin lymphomas that are infected with Epstein-Barr virus (EBV). EBV is found in cancer cells of up to half of all patients with Hodgkin and non-Hodgkin lymphoma. This suggests that it may play a role in causing lymphoma. The cancer cells infected by EBV are able to hide from the body's immune system and escape being killed. The investigators previously tested whether special white blood cells (called T cells) that were trained to kill EBV-infected cells could affect these tumors, and in many patients the investigators found that giving these trained T cells caused a complete or partial response.

Other cancers express specific proteins that can be targeted in the same way. The investigators have been able to infuse such tumor-targeted cells into up to 10 patients with lymphoma who do not have EBV, and seen some complete responses. Importantly, the treatment appears to be safe. Therefore, the investigators now want to test whether the investigators can direct these special T cells against other types of cancers that carry similar proteins called tumor-associated antigens (TAAs). These proteins are specific to the leukemia cell, so they either do not show up, or show up in low quantities, on normal human cells.

The investigators will grow T cells from patients' stem cell donors in the laboratory in a way that will train them to recognize the tumor proteins WT1, PRAME and Survivin, which are expressed on most ALL cancer cells. The cells will be infused at least 30 days post-allogeneic HSCT. In this study, the investigators want to see whether these cells will be able to recognize and kill leukemia cells that express these antigens. These donor-derived multiTAA-specific T cells are an investigational product not yet approved by the U.S. Food and Drug Administration.

The purpose of this study is to find the largest safe dose of donor-derived multiTAA-specific T cells for patients with ALL.

DETAILED DESCRIPTION:
To make donor-derived multiTAA-specific T cells, the investigators will collect blood from the patient's stem cell donor, and mix the donor's T cells with small pieces of the tumor proteins WT1, PRAME and Survivin. These protein fragments stimulate the donor T cells to grow and react against these proteins in such a way that they will recognize and kill cancer cells that express these proteins. Once sufficient numbers of multiTAA-specific T cells have been made, the investigators test them to make sure they target the patient's cancer cells, but not their normal healthy cells.

The multiTAA-specific T cells will be administered as a single intravenous (IV) infusion over 10 minutes. The patient's cancer will be assessed within 4 weeks prior to the T cell infusion, at 4-6 weeks, and again at 8-12 weeks after the infusion. If at least 4 weeks after the infusion there is no change or a reduction in the number of cancer cells measured in the bone marrow, or a decline in cancer-specific markers in the blood, patients may receive up to six (6) additional doses of the T cells at least 4 weeks apart. All of the treatments will be given by the Center for Cell and Gene Therapy at Houston Methodist Hospital or Texas Children's Hospital.

For at least 4 weeks after the infusion, patients may not receive any other anti-cancer treatments, such as radiation therapy or chemotherapy, with the exception of drugs like dasatinib. Patients who do receive any other therapies will be taken off treatment, and will not be able to receive additional doses of T cells.

This is a dose escalation study, which means that at the beginning, patients will be started on the lowest dose (1 of 3 different levels) of T cells. Once that dose level proves safe, the next group of patients will be started at the next highest dose. This process will continue until all 3 dose levels have been studied. If side-effects are too severe, the dose will be lowered or the T cell injections will be stopped.

Before being treated, patients will undergo a series of standard medical tests:

* Physical exam.
* Blood tests to measure blood cells, kidney and liver function.
* Measurement of ALL (done by a bone marrow biopsy or blood tests).
* Pregnancy test, if patient is a female who can have children.

Patients will undergo standard medical tests both during the T cell infusions and after:

* Blood tests to measure blood cells, kidney and liver function.
* Measurement of disease 4-6 weeks and 8-12 weeks after the T cell infusion (done by bone marrow biopsy or blood tests).

Active participation in this study will last for approximately one (1) year. If the patient receives additional doses of the T cells as described above, their active participation will last until one (1) year after the last dose of T cells. We will then contact the patient once a year for up to 4 additional years (total of 5 years follow-up) in order to evaluate disease response long-term.

ELIGIBILITY:
Inclusion Criteria:

Only patients who receive infusions in the integrated Cell and Gene Therapy (CAGT) Transplant program at Texas Children's Hospital (TCH) or Houston Methodist Hospital (HMH) are eligible for this study.

1. Patients will be eligible to receive donor-derived multiTAA-specific T cells following any type of allogeneic HSCT as:

   (i) Adjuvant therapy for ALL (Group A), or (ii) Treatment for relapsed/residual ALL disease (Group B)

   Residual disease at the time of transplant or post-transplant relapse is defined as PCR positivity, specific cytogenetic abnormalities, an abnormal population on flow cytometry, or increased blasts on bone marrow biopsy or in the peripheral blood. Minimal residual disease (MRD )will be defined as detection in blood or marrow of any of the following:

   (i) Any leukemia-specific marker (such as t(12;21); t(9;22) or t(4;11)) documented in the patient's leukemia cells pre-transplant on a post-transplant evaluation.

   (ii) A leukemia-specific phenotype (e.g. expression of markers including CD10 and/or CD19 or CD3 and/or CD4 or CD8) post-transplant at a level greater than or equal to 0.01%.

   (iii) Mixed donor chimerism (greater than 20%).
2. Life expectancy greater than or equal to 6 weeks.
3. Karnofsky/Lansky score of greater than or equal to 50.
4. Patient or parent/guardian capable of providing informed consent.
5. Bilirubin less than or equal to 2X upper limit of normal.
6. AST less than or equal to 3X upper limit of normal.
7. Serum creatinine less than or equal to 2X upper limit of normal.
8. Hgb greater than or equal to 7.0 g/dL (can be transfused).
9. Pulse oximetry of greater than 90% on room air.
10. Sexually active patients must be willing to utilize one of the more effective birth control methods for 6 months after the ATL infusion. Male partner should use a condom.
11. Available donor-derived multiTAA-specific T cell line.
12. No other investigational anti-neoplastic therapy for one month prior to entry in this study.
13. Undergoing Stem Cell Transplant at CAGT

Exclusion Criteria:

1. Patients receiving ATG or Campath within 28 days of infusion.
2. Patients receiving a Donor Lymphocyte Infusion (DLI) within 4 weeks of planned T cell infusion.
3. Less than 30 days post-allogeneic stem cell transplant.
4. Severe intercurrent infection.
5. Evidence of GVHD greater than Grade II.
6. Pregnant or lactating.
7. Currently taking corticosteroids (greater than 0.5 mg/kg/day prednisone or equivalent).

Donor Eligibility:

Donors for allogeneic (i.e. HLA matched or mismatched related or unrelated) stem cell transplants who have fulfilled eligibility for and consented to stem cell donation as per the stem cell transplant program's standard operating procedures. Subjects must be at least 12 kg or 24 pounds to be eligible for stem cell donation. The stem cell donor will have already been selected by the primary Bone Marrow Transplant attending according to CAGT SOPs for Donor Evaluation, Donor Selection, and Donor Deferral. If a donor has been chosen for the transplant based on urgent medical need, that same donor will also be used for T cell generation, provided that there are no new reasons for ineligibility since the stem cell collection. In this study, the subject's hematopoietic stem cell donor will also be the donor for the T cells.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02; Primary Completion 2019-10-29 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicities (DLTs). | 4 weeks
  Maximum tolerated dose (MTD) of multiTAA-specific T cells among the three pre-specified dose levels.

SECONDARY OUTCOMES:
Number of patients with a decrease in the marker of disease. | 4 weeks
  To obtain information on the anti-tumor effects of adoptively transferred donor-derived multiTAA-specific T cells in patients with ALL.
Median number of T cells post-infusion. | 1 year
  To obtain information on the expansion and persistence of adoptively transferred donor-derived multiTAA-specific T cells in patients with ALL.

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Omer, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

DOCUMENTS (1):
  • Informed Consent Form (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT02475707/ICF_000.pdf